CLINICAL TRIAL: NCT05651373
Title: The Clinical Features and Pregnancy Outcomes of Patients With Rheumatoid Arthritis :a Prospective Cohort Study
Brief Title: The Clinical Features and Pregnancy Outcomes of RA Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Qiang Shu, Chief Physician, Qilu Hospital of Shandong University
Other Study IDs: RA with Pregnancy QiluH
Record Dates: First submitted 2022-11-15; First posted 2022-12-15 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Rheumatoid Arthritis; Pregnancy Related
Keywords: Rheumatoid Arthritis; Pregnancy outcomes; Clinical features; Risk factors
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Prednisone; prednylidene; Hydroxychloroquine; Certolizumab Pegol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Early, intermediate and late peripheral blood specimens、cord blood specimens、placental tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients not using TNF inhibitors(TNFi): The cohort includes the RA patients in pregnancy.
  Drug: Hydroxychloroquine(HCQ)，200mg, po, twice per day (Bid) prescribed at the beginning and adjusted due to patient response.
  Drug: Prednisone(Pred)，5-30mg, po, once per day (qd) prescribed at the beginning and adjusted due to patient response.
  Interventions: Drug: Prednisone; Drug: Hydroxychloroquine
- patients using TNF inhibitor (TNFi): The cohort includes the RA patients in pregnancy.
  Drug: Hydroxychloroquine(HCQ)，200mg, po, twice per day (Bid) prescribed at the beginning and adjusted due to patient response.
  Drug: Prednisone(Pred)，5-30mg, po, once per day (qd) prescribed at the beginning and adjusted due to patient response.
  Drug: TNFi ,such as Certolizumab Pegol (Cimzia)，200mg, iH,q2w, once two weeks (q2w) prescribed from the beginning and adjusted due to patient response.
  Interventions: Drug: Prednisone; Drug: Hydroxychloroquine; Drug: CertolizumabPegol injection

INTERVENTIONS:
Drug: Prednisone — 5-30mg, po, once per day(Qd) prescribed if needed and adjusted due to patient response
  Other Names: Pred
Drug: Hydroxychloroquine — 200mg, po, twice per day (Bid) prescribed if needed and adjusted due to patient response.
  Other Names: HCQ
Drug: CertolizumabPegol injection — 200mg, iH,q2w, once two weeks (q2w) prescribed from the beginning and adjusted due to patient response.
  Other Names: Cimzia
  Groups: patients using TNF inhibitor (TNFi)

SUMMARY:
This study includes RA patients in pregnancy, who are using different treatment regimens，including prednisone, hydroxychloroquine, and/or TNF inhibitors. The maternal disease activity, pregnancy outcomes, maternal and fetal safety are assessing during the trimester of pregnancy. The effects of different therapies and risk factors for adverse pregnancy outcomes will be analysis.

DETAILED DESCRIPTION:
To study the risk factors of poor pregnancy outcomes in RA patients, and evaluate impact of different therapies on the maternal and fetal health.

The follow-up study will be scheduled every 4 weeks from confirmed pregnancy until delivery, records the disease activity of RA, pregnancy outcome and safety with the help of the "smart disease management system (SSDM)" and face-to-face consultations.

The effects of different therapies on maternal and fetal will be valued

ELIGIBILITY:
Inclusion Criteria:

- 1.Age between 20 and 45 years old.

2.Diagnosis of RA: Approved by the American College of Rheumatology and the European League Against Rheumatism in 2010.

Involved joints 1 large joint (0 points) 2-10 large joints (1 point) 1-3 small joints (with or without large joints) (2 points) 4-10 small joints (with or without large joints) (3 points) more than 10 small joints (at least one small joint) (5 points)

Serological indicators RF and ACPA negative (0 points) RF and ACPA, at least one of which is low titer positive. (2 points) RF and ACPA with at least one high titer positive (3 points)

Acute chronotropic reactants Both CRP and ESR normal (0 points) Abnormal CRP or ESR (1 point)

Duration of synovitis <6 weeks (0 points)

≥6 weeks (1 point)

3.Voluntary participation in this study, willingness to administer medication and follow up according to the treatment plan, and signing of an informed consent form.

Exclusion Criteria:

* Women who meet any of the following criteria will be excluded from the study

  1. Any known etiology of previous pregnancy loss

     1. Known paternal, maternal or embryonic chromosomal abnormalities.
     2. Maternal endocrine dysfunction: luteal insufficiency; polycystic ovary syndrome; premature ovarian failure (follicular phase stimulating hormone, FSH ≥ 20uU/L).
     3. Hyperprolactinemia; diabetes mellitus; other abnormalities of the hypothalamic pituitary-adrenal axis.
     4. Maternal anatomical abnormalities: uterine malformations; Asherman syndrome; cervical insufficiency; uterine fibrosis greater than 5 cm. vaginal infection.
     5. Any known serious cardiac, hepatic, renal, hematologic or endocrine disease.
  2. Any active infection, including bacterial, alisla virus (VZV), human immunodeficiency virus (HIV), human papillomavirus (HPV), syphilis, tuberculosis, fungal infections, etc.
  3. Hypersensitivity to prednisone, hydroxychloroquine, low molecular weight heparin or aspirin
  4. History of the following diseases.

     1. Past history of peptic ulcer or upper gastrointestinal bleeding.
     2. Past history of malignancy.
     3. Past history of epilepsy or mental disorder.
     4. Female has been diagnosed with SLE
     5. Women who do not consent or are unable to complete pregnancy and postpartum follow-up.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: female with pregnance in accordance with the diagnostic criteria of Rheumatoid arthritis in 2010.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-07-30 (Actual); Primary Completion 2023-08-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The percentage of patients who achieve clinical remission using DAS28-CRP | through study completion, an average of 10 months
  The percentage of patients whose DAS28 achieve remission（DAS28-CRP≤ 2.6）and Low Disease Activity (DAS28-CRP ≤3.2) .

SECONDARY OUTCOMES:
Early fetal loss | within 10 weeks of gestation
  Spontaneous pregnancy loss within 10 weeks of gestation
Late fetal loss | after 10 weeks of gestation
  Spontaneous pregnancy loss after 10 weeks of gestation
Still birth | after 10 weeks of gestation
  Spontaneous pregnancy loss after 10 weeks of gestation.
Preterm delivery | between 28 and 37 weeks of gestation
  Live birth before 37 weeks of gestation.
Low-weight birth | after 28 weeks of gestation
  newborns with low weight (<2500g)
Premature rupture of membranes | after 28 weeks of gestation
  the number of participants complicated with placental abruption
Placental abruption | after 28 weeks of gestation
  the number of participants complicated with placental abruption
Fetal growth retardation (FGR) | after 12 weeks of gestation
  weight below the 10th percentile for the gestational age
Number of participants with low amniotic fluid during pregnancy | after 12 weeks of gestation
  the number of participants whose B-ultrasound indicates low amniotic fluid during pregnancy
Number of participants with abnormal S / D values during pregnancy | after 12 weeks of gestation
  the number of participants whose B-ultrasound indicates abnormal S / D values during pregnancy
Number of participants with placental hematoma during pregnancy | during pregnancy
  the number of participants whose B-ultrasound indicates placental hematoma during pregnancy
Eclampsia | after 20 weeks of gestation
  New-onset hypertension after 20 weeks of gestation, with or without proteinuria > 300mg/24h, with or without any organ damage with seizures
Gestational diabetes | through study completion, an average of 10 months
  the number of participants who were diagnosed with gestational diabetes
Gestational hypertension | through study completion, an average of 10 months
  the number of participants who were diagnosed with gestational hypertension
Number of participants with placental infarction | at delivery
  the number of participants whose placenta with infarction.
Change From Baseline in C-reactive Protein (CRP) | through study completion, an average of 10 months
  Change from Baseline in C-reactive Protein (CRP), CRP will be measured with blood samples.
Erythrocyte Sedimentation Rate (ESR) | through study completion, an average of 10 months
  Change from Baseline in Erythrocyte Sedimentation Rate (ESR), ESR will be measured with blood samples.
Live birth rate | After 28 weeks of gestation
  Percentage of all patients that lead to live birth after 28 weeks of gestation
Change from baseline Simplified Disease Activity Index (SDAI) | through study completion, an average of 10 months
  SDAI score exceeding 26 is considered high disease activity; 11 <SDAI ≤26，moderate disease activity; 3.3 <SDAI ≤11, low disease activity; remission is SDAI score ≤ 3.3.
Change from baseline Clinical Disease Activity Index (CDAI) | through study completion, an average of 10 months
  CDAI > 22 is considered high disease activity; 10 <CDAI ≤ 22, moderate disease activity; 2.8 <CDAI ≤10, low disease activity; remission is CDAI score ≤2.8.
swollen joint number (SW28) | through study completion, an average of 10 months
  SW28 means the number of joints with swelling counted in 28 synovial joints, including proximal interphalangeal joints (10 joints), metacarpophalangeal joints (10), wrists (2), elbows (2), shoulders (2) and knees (2) bilateral.
tenderness joint number (T28) | through study completion, an average of 10 months
  T28 means the number of joints with tenderness upon touching counted in 28 synovial joints, including proximal interphalangeal joints (10 joints), metacarpophalangeal joints (10), wrists (2), elbows (2), shoulders (2) and knees (2) bilateral.
patient global assessment(PGA) | through study completion, an average of 10 months
  patient global assessment(PGA)
Health Assessment Questionnaire (HAQ) | through study completion, an average of 10 months
  Health Assessment Questionnaire (HAQ)
Percentage of patients achieving Boolean remission | through study completion, an average of 10 months
  Clinical remission was defined when the number of swollen joints ≤1, the number of painful joints ≤1, CRP ≤1 mg/dl and the patient's overall score of the disease ≤1 were also satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoyun Yang, Study Director — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No